CLINICAL TRIAL: NCT03717064
Title: An Open-Label, Fixed Sequence, Two-Period Study to Investigate the Effect of RO7049389 on the Pharmacokinetics of Pitavastatin in Healthy Volunteers
Brief Title: A Study to Investigate the Effect of RO7049389 on the Pharmacokinetics of Pitavastatin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YP40218
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Results first posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2019-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — pitavastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pitavastatin (Experimental): Period 1: Participants will receive a single dose of pitavastatin on Day 1, followed by a wash-out period of at least 7 and up to 21 days.
  Period 2: Participants will receive RO7049389 on Days 1-6. Participants will also receive a single dose of pitavastatin on Day 4.
  Interventions: Drug: RO7049389; Drug: Pitavastatin

INTERVENTIONS:
Drug: RO7049389 — RO7049389 will be taken orally, in tablet form, BID on Days 1-6 of Period 2.
Drug: Pitavastatin — Pitavastatin will be taken orally, in tablet form, once on Day 1 of Period 1, and once on Day 4 of Period 2.

SUMMARY:
The main purpose of the study is to characterize the interaction between RO7049389 and the cholesterol-lowering drug, pitavastatin, in healthy volunteers. There is no intended clinical benefit to this study. The total duration of the study for each participant is approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria

* Healthy, as judged by the Investigator. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, and based on the laboratory safety test results at screening and Day -1
* Body mass index (BMI) between 18 to 30 kg/m2 (inclusive) at screening
* Female participants: 1) Must be either surgically sterile (by means of hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy) or post-menopausal for at least one year (defined as amenorrhea >/=12 consecutive months without another cause, and confirmed by follicle-stimulating hormone (FSH) level. 2) Participants must not be pregnant or lactating.
* Male participants: 1) Female partners must not be pregnant or lactating. 2) Must agree to remain abstinent (refrain from heterosexual intercourse) or must agree to use a condom with spermicide during the treatment period and for at least 28 days after the last dose of study drug with female partners of childbearing potential. 3) Must agree to refrain from donating sperm during the treatment period and for at least 28 days after the last dose of study drug

Exclusion Criteria

* Have a history or symptoms of any clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, oncologic or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study treatment; or of interfering with the interpretation of data
* Confirmed (based on the average of 3 separate resting BP measurements in a supine position, after at least 5 minutes rest) systolic BP greater than 140 or less than 90 mmHg, and diastolic BP greater than 90 or less than 50 mmHg at screening and Day -1
* Personal history or family history of congenital long QT syndrome and/or cardiac sudden death
* History of Gilbert's syndrome
* Participants who have had significant acute infection, e.g., influenza, local infection, acute gastrointestinal symptoms or any other clinically significant illness within two weeks of dose administration
* Any confirmed significant allergic reactions (urticaria or anaphylaxis) against any drug, or multiple drug allergies (non-active hay fever is acceptable)
* Taking any herbal medications or substances (e.g., tea) or supplements (including vitamins), or traditional Chinese medicines (TCM) or over-the-counter (OTC) medications within 14 days of first dosing or within 5 times the elimination half-life of the medication prior to first dosing, whichever is longer
* History of having received any systemic anti-neoplastic (including radiation) or immunemodulatory treatment (including systemic oral or inhaled corticosteroids) </=6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study
* Are currently enrolled in or have participated in any other clinical study involving an investigational product or in any other type of medical research within the last 30 days or 5 half lives (whichever is longer)
* Donation or loss of blood or blood products in excess of 500 mL within 3 months of screening and for the duration of the study
* Positive test for drugs of abuse (including recreational drugs) and/or positive alcohol test and/or positive cotinine test at screening and on Day -1
* Positive test at screening of any of the following: Hepatitis A virus (HAV IgM Ab), hepatitis B virus (HBsAg or HBcAb), hepatitis C virus (HCV RNA or HCV Ab) or human immunodeficiency virus (HIV-1 and HIV-2 Ab)
* History of alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink = 10 grams of alcohol) and/or drug abuse within 12 months of screening
* Use of >5 cigarettes or equivalent nicotine-containing product per day prior to screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-LaRoche
Locations (1):
- Covance Research Unit - Daytona, Daytona Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited healthy adult participants at one site in the United States.
Pre-assignment Details: This study had two periods. Period 1: Participants received a single dose of pitavastatin, followed by a washout period of 7-21 days. Period 2: Participants received a single dose of pitavastatin along with a twice-daily dose of RO7049389.
Groups:
- Pitavastatin/RO7049389: Period 1: Participants received a single dose of pitavastatin on Day 1, followed by a wash-out period of at least 7 days and up to 21 days.
  Period 2: Participants received RO7049389 on Days 1-6. Participants also received a single dose of pitavastatin on Day 4.
Period: Period 1
Arm/Group | Pitavastatin/RO7049389
Started | 18
Completed | 18
Not Completed | 0
Period: Period 2
Arm/Group | Pitavastatin/RO7049389
Started | 18
Completed | 17
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.2 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Period 1: Maximum Plasma Concentration (Cmax) of Pitavastatin
Time Frame: Period 1 Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
ng/mL | 23.8 (42.7)

2. Primary Outcome: Period 1: Plasma Concentration Versus Time (Area Under the Curve, AUC0-inf) of Pitavastatin
Time Frame: Period 1 Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
h*ng/mL | 78.6 (41)

3. Primary Outcome: Period 1: Time to Maximum Concentration (Tmax) of Pitavastatin
Time Frame: Period 1 Day 1
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
hours (h) | 1.5 [0.5 to 2]

4. Primary Outcome: Period 1: Apparent Total Clearance (CL/F) of Pitavastatin
Time Frame: Period 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
L/h | 25.4 (39.9)

5. Primary Outcome: Period 1: Volume of Distribution (V/F) of Pitavastatin
Time Frame: Period 1 Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
Liters (L) | 525 (41.3)

6. Primary Outcome: Period 1: Elimination Half-Life (T1/2) of Pitavastatin
Time Frame: Period 1 Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
h | 14.3 (32.4)

7. Primary Outcome: Period 2: Maximum Plasma Concentration (Cmax) of Pitavastatin
Time Frame: Period 2 Day 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
ng/mL | 33.5 (52.7)

8. Primary Outcome: Period 2: Plasma Concentration Versus Time (Area Under the Curve, AUC0-inf) of Pitavastatin
Time Frame: Period 2 Day 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
h*ng/mL | 129 (50.7)

9. Primary Outcome: Period 2: Time to Maximum Concentration (Tmax) of Pitavastatin
Time Frame: Period 2 Day 4
Measure: Median (Full Range); unit: h
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
h | 2 [0.5 to 4]

10. Primary Outcome: Period 2: Apparent Total Clearance (CL/F) of Pitavastatin
Time Frame: Period 2 Day 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
L/h | 15.6 (45)

11. Primary Outcome: Period 2: Volume of Distribution (V/F) of Pitavastatin
Time Frame: Period 2 Day 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
L | 220 (59.3)

12. Primary Outcome: Period 2: Elimination Half-Life (T1/2) of Pitavastatin
Time Frame: Period 2 Day 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
h | 9.78 (49)

13. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: From the start of Period 1 through safety follow-up (Period 2, Day 34)
Measure: Number; unit: Percentage of Participants
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 18
Percentage of Participants | 39

14. Secondary Outcome: Period 2: Cmax of RO7049389
Time Frame: Period 2 Days 3-4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
ng/mL
  RO7049389 | 15400 (58.1)
  RO7049389 + Pitavastatin | 17600 (48.4)

15. Secondary Outcome: Period 2: AUC-tau of RO7049389
Time Frame: Period 2 Days 3-4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
h*ng/mL
  RO7049389 | 62700 (92.8)
  RO7049389 + Pitavastatin | 68500 (81.8)

16. Secondary Outcome: Period 1: Cmax of Pitavastatin Lactone
Time Frame: Period 1 Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
ng/mL | 14.4 (23.5)

17. Secondary Outcome: Period 1: AUC0-inf of Pitavastatin Lactone
Time Frame: Period 1 Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
h*ng/mL | 193 (27.4)

18. Secondary Outcome: Period 1: AUC Ratio of Pitavastatin Lactone to Pitavastatin
Time Frame: Period 1 Day 1
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
Ratio | 2.45 [2.17 to 2.78]

19. Secondary Outcome: Period 2: Cmax of Pitavastatin Lactone
Time Frame: Period 2 Day 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
ng/mL | 6.39 (24.4)

20. Secondary Outcome: Period 2: AUC0-inf of Pitavastatin Lactone
Time Frame: Period 2 Day 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
h*ng/mL | 81.7 (19.9)

21. Secondary Outcome: Period 2: AUC Ratio of Pitavastatin Lactone to Pitavastatin
Time Frame: Period 2 Day 4
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Pitavastatin/RO7049389
Number analyzed (Participants) | 17
Ratio | 0.636 [0.504 to 0.802]

ADVERSE EVENTS:
Time Frame: From the start of Period 1 through safety follow-up (Period 2, Day 34)
Arm/Group | Pitavastatin/RO7049389
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 7/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pitavastatin/RO7049389 (N=18)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT03717064/Prot_SAP_000.pdf